CLINICAL TRIAL: NCT00533091
Title: A Phase 1B, Randomized, Double-blind, Placebo-Controlled, Multicenter Study to Evaluate Safety of Multiple-Dose, Intravenously Administered MEDI-545, A Fully Human Anti Interferon-Alpha Monoclonal Antibody, In Adult Patients With Dermatomyositis or Polymyositis
Brief Title: A Study to Evaluate Safety of Multi-Dose MEDI-545 in Adult Patients With Dermatomyositis or Polymyositis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP151
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: DERMATOMYOSITIS OR POLYMYOSITIS
MeSH Terms: conditions — Dermatomyositis | interventions — sifalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): MEDI-545
  Interventions: Biological: MEDI-545
- 2 (Other): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MEDI-545 — MEDI-545 is supplied as a sterile liquid containing 0.75 mL of MEDI-545 solution at a concentration of 100 mg/mL in a 3 mL single-use glass vial.
  Dosage, frequency and duration: MEDI-545 (0.3, 1.0, 3.0, or 10.0 mg/kg) will be administered via infusion over at least 60 minutes every 2 weeks for 26 weeks.
  Arms: 1
Other: Placebo — Dosage form: Placebo is supplied as a sterile liquid containing a 0.75 mL solution in a 3 mL single-use vial.
  Dosage, frequency and duration: Placebo (0.3, 1.0, 3.0, or 10.0 mg/kg) will be administered via infusion over at least 60 minutes every 2 weeks for 12 weeks.
  Thereafter, subjects will receive MEDI-545, at the dose specified in the dose cohort they are assigned, every 2 weeks for an additional 12 weeks.
  Arms: 2

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of multiple IV doses of MEDI-545 in adult patients with myositis.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the safety and tolerability of multiple intravenous (IV) doses of MEDI-545 in adult patients with dermatomyositis (DM) or polymyositis (PM).

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults at least 18 years of age at the time of randomization;
* Written informed consent obtained from the patient or the patient's legal representative prior to receipt of any study medication or beginning study procedures;
* Probable or definite PM or DM according to the Bohan and Peter criteria (Bohan, 1975);
* For patients with PM, documentation of a muscle biopsy result that is consistent with the diagnosis of PM;
* All patients including those with DM must meet at least two of the following criteria:
* Strength in MMT greater ≥ 80/150 but ≤ 125/150 using the MMT-8 muscle group testing;
* Patient Global Activity Assessment by visual analog scale (VAS)≥ 2.0 cm on a 10 cm scale, which is included as part of CLINHAQ;
* Physician Global Activity Assessment by VAS ≥ 2.0 cm on a 10 cm scale, which is included as part of MDAAT;
* CLINHAQ disability index ≥ 0.25;
* Global extramuscular activity assessment ≥ 1.0 cm on a 10-cm VAS scale (this measure is the physician's composite evaluation and is based on assessments of activity scores on the constitutional, cutaneous, skeletal, gastrointestinal, pulmonary and cardiovascular scales of the MDAAT;
* Subjects with PM must have an elevation of serum CK or aldolase at a minimum level of 1.3 x upper limit of normal (ULN) or serum CK or aldolase at least 2-fold higher than the patient's own lowest value since diagnosis;
* Subjects with DM must have either an elevated CK or aldolase as above (per inclusion criterion #6) or other laboratory evidence of active myositis. This could include either abnormal signal on skeletal muscle MRI suggestive of inflammation or an electromyogram demonstrated muscle membrane irritability (e.g., fibrillation potentials, positive sharp waves, complex repetitive discharges) and short duration, small amplitude, polyphasic motor unit action potentials;
* For patients randomized to Dose Cohorts 1.2, 3A and 4: median fold overexpression of the top 25 type I IFN inducible genes of four-fold or greater in whole blood at the time of screening; For patients randomized to dose cohort 3B: low or negative expression of type I IFN-inducible genes;
* Sexually active women, unless surgically sterile (including tubal ligation) or at least 2 years postmenopausal, must use an effective method of avoiding pregnancy (including oral, injectable, transdermal, or implanted contraceptives, intrauterine device, diaphragm with spermicide, cervical cap, abstinence, and sterile sexual partner) in addition to the use of condoms (male or female condoms with spermicide) from screening through end of study. Cessation of birth control after this point should be discussed with a responsible physician. Sexually active males, unless surgically sterile, must likewise practice two effective methods of birth control (condom with spermicide or abstinence) and must use such precautions from Study Day 0 through end of study;
* Ability to complete the study period, including follow-up period, of up to 350 days; and
* Willing to forego other forms of experimental treatment during the study.

Exclusion Criteria:

* Receipt of MEDI-545 in any previous clinical study or prior randomization into the trial;
* History of allergy or reaction to any component of the study drug formulation;
* Inclusion body myositis, cancer-associated myositis, myositis associated with another connective tissue disease, environmentally-associated myositis, or drug-related myopathy;
* A history of or a family history of noninflammatory myopathy, scapular winging, atrophy, or hypertrophy of the calf muscles;
* Receiving prednisone > 35 mg/day (or an equivalent dose of another corticosteroid) within 14 days before Study Day 0;
* Receiving the following dosages of medications within 28 days before Study Day 0: hydroxychloroquine > 600 mg/day, mycophenolate mofetil > 3 g/day, methotrexate > 25 mg/week, azathioprine > 3 mg/kg/day, or any dose of cyclophosphamide, cyclosporine, or thalidomide;
* Have received fluctuating doses of antimalarials, mycophenolate mofetil, methotrexate, leflunomide, or azathioprine within 28 days before Study Day 0 or fluctuating doses of corticosteroids within 14 days before Study Day 0;
* Have received leflunomide > 20 mg/day in the 6 months prior to Study Day 0;
* Treatment with any investigational drug therapy within 28 days before Study Day 0 or biologic therapies (eg, rituximab) within 30 days or 5 half-lives of the biologic agent, whichever is longer, before Study Day 0;
* In the investigator's opinion, evidence of clinically significant active infection, including ongoing, chronic infection, within 28 days before Study Day 0;
* A history of severe viral infection as judged by the investigators, including severe infections of either CMV or the herpes family such as disseminated herpes, herpes encephalitis, ophthalmic herpes;
* Herpes zoster ≤ 3 months prior to Study Day 0;
* Evidence of infection with hepatitis B or C virus or HIV-1 or HIV-2, or active infection with hepatitis A, as determined by results of testing at screening;
* Vaccination with live attenuated viruses within 28 days before Study Day 0;
* Pregnancy (sexually active women, unless surgically sterile or at least 2 years post-menopausal, must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to study drug administration on Study Day 0);
* Breastfeeding or lactating women;
* History of alcohol or drug abuse < 1 year prior to Study Day 0;
* History of cancer, except for basal cell carcinoma or carcinoma in situ of the cervix treated with apparent success with curative therapy more than 1 year prior to Study Day 0;
* History of active tuberculous infection;
* History of latent tuberculous infection or newly positive TB skin test (reaction defined as ≥ 10 mm in diameter if not on systemic immunosuppressive medication or ≥ 5 mm if on systemic immunosuppressive medication) without completion of an appropriate course of treatment or ongoing prophylactic therapy;
* A history of coagulation disorders that in the opinion of the investigator would contraindicate skin or muscle biopsies;
* Elective surgery planned from the time of screening through Study Day 196;
* At screening blood tests (must be within 28days before Study Day 0) any of the following:

  * Serum creatinine > 4.0 mg/dL,
  * Neutrophils < 1,500/mm3,
  * Platelet count < 50,000/mm3;
* History of any disease, evidence of any current disease (other than DM or PM), any finding upon physical examination, or any laboratory abnormality, that, in the opinion of the investigator or medical monitor, may compromise the safety of the patient in the study or confound the analysis of the study; or
* Any employee of the research site who is involved with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-04; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoints of the study are safety and tolerability of multiple intravenous (IV) doses of MEDI-545 in adult patients with Dermatomyositis or Polymyositis, assessed primarily by summarizing AEs assessing changes in viral cultures and titers. | 12 months

SECONDARY OUTCOMES:
The secondary endpoints of the study are the PK and IM of multiple IV doses of MEDI-545. | 12 months
The third endpoint of the study are the evaluations of disease activities. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Ethgen, M.D., Study Director — MedImmune LLC
Locations (14):
- United States (14):
  - Research Site, Scottsdale, Arizona
  - Research Site, Stanford, California
  - Research Site, Whittier, California
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Miami, Florida
  - Research Site, Evansville, Indiana
  - Research Site, Kansas City, Kansas
  - Research Site, Baltimore, Maryland
  - Research Site, Cumberland, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Lebanon, New Hampshire
  - Research Site, Lake Success, New York
  - Research Site, Portland, Oregon
  - Research Site, Duncansville, Pennsylvania

REFERENCES:
- [Derived] Higgs BW, Zhu W, Morehouse C, White WI, Brohawn P, Guo X, Rebelatto M, Le C, Amato A, Fiorentino D, Greenberg SA, Drappa J, Richman L, Greth W, Jallal B, Yao Y. A phase 1b clinical trial evaluating sifalimumab, an anti-IFN-alpha monoclonal antibody, shows target neutralisation of a type I IFN signature in blood of dermatomyositis and polymyositis patients. Ann Rheum Dis. 2014 Jan;73(1):256-62. doi: 10.1136/annrheumdis-2012-202794. Epub 2013 Feb 23. PMID 23434567